CLINICAL TRIAL: NCT05362513
Title: Comparative Study Between Topical Permethrin 5% and Oral Ivermectin for the Treatment of Scabies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Naheed khan, principal investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHatd-ETH-23-derm-22; 131/CPSP (Other: CPSP)
Record Dates: First submitted 2022-04-21; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Scabies
Keywords: Permethrin 5%; scabies; ivermectin
MeSH Terms: conditions — Scabies | interventions — Ivermectin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A(permethrin topical) (Active Comparator): Group A received Permethrin 5% twice with a one-week interval, whereas Group B received a single dose of oral ivermectin 200 mcg per kg.
  Interventions: Drug: Permethrin Cream
- Group B oral ivermectin (Active Comparator): Group A received Permethrin 5% twice with a one-week interval, whereas Group B received a single dose of oral ivermectin 200 mcg per kg
  Interventions: Drug: Ivermectin Tablets

INTERVENTIONS:
Drug: Ivermectin Tablets — Group B received a single dose of oral ivermectin 200 mcg per kg
  Arms: Group B oral ivermectin
Drug: Permethrin Cream — Group A received Permethrin 5% twice with a one-week interval.
  Arms: Group A(permethrin topical)

SUMMARY:
Globally, Scabies infects 300m people each year. In children of developing countries, its prevalence is expected to be about 5 to 10%.In Pakistan, Scabies accounts for 38% of dermatological diseases. Males were more prone to infestation than females, and early school-aged children were the most vulnerable. It was more widespread in urban than in rural areas. A distinct seasonal pattern emerged, with the biggest infestation occurring in the winter and the lowest in the summer. Scabies risk factors estimated 89% of the variation in its prevalence.

The classic scabies symptoms include an erythematous papular eruption, burrows, and intense itching. It is usually transmitted by prolonged skin-skin contact. Predilection sites are fingers, axilla, elbows, waist, belly, groin, genital area, etc. Classic scabies can be diagnosed by proper taking history and clinical symptoms. Some of the clinical variations of scabies are Crusted, nodular, and bullous. On examination under a microscope of scrapings collected from skin lesions, finding the mites, eggs, confirms the infestation of scabies .

Topical permethrin and oral ivermectin are the medications of choice for scabies mite elimination. Topical Permethrin 5% applied for 9-14 hours for adults than for children only 8-9 hours. Permethrin 5% only single dose is enough but the second dose can be applied after an interval of 2 weeks if the etiology is still there. Ivermectin is now used to treat scabies, with an effective dosage of 150 to 200 μg/kg given once or may give twice after interval of two weeks. The positives include a single dosage and improved compliance in resistant infestations and situations where head-to-toe topical administration is logistically problematic, such as huge outbreaks or mentally impaired individuals. Fever, arthralgia, myalgia, dizziness, headache, hypotension, tachycardia, and lymphadenopathy have all been reported as adverse effects. There have also been reports of a prolonged prothrombin time, a transient EKG, and variations in liver enzymes.

The study's implications are to analyze the safety and efficacy of these two drugs in order to better treat patients with evidence-based management and rule out any potential adverse effects.

DETAILED DESCRIPTION:
A randomized controlled trial study (single-blind) was done In the Dermatology Unit of the CMH, Abbottabad from June to November 2021 after Ethical Review Board approval, the 100 patients aged 5-80 years after informed consent were enrolled using a technique of non-probability consecutive sampling. The sample size for two proportions was determined using the WHO sample size calculator, with a threshold of significance of 5%. The anticipated population proportion P1 was 80%, while the anticipated population proportion P2 was 46.6% 12. The sample size was calculated to be 100.

ELIGIBILITY:
Inclusion Criteria:

* More than 2 years
* More than 15kg of body weight
* attended the Dermatology department

Exclusion Criteria:

* Patients under the age of two years
* pregnant
* breastfeeding women
* those with a background of seizures, severe symptoms of systemic illnesses,
* immunosuppression diseases,
* Norwegian scabies
* those who had taken any topical or systemic acaricide medication for one month before the trial

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Complete clearance (outcome assessment at 7 and 14 days post initiation of treatment) | 2 weeks
  For randomization, the final recruited 100 participants (57 females and 43 men; mean+SD age 35.28+18.51 years, range 5 to 80), randomly assigned to one of two groups i.e. Group A received Permethrin 5% twice with a one-week interval, whereas Group B received a single dose of oral ivermectin 200 mcg per kg. They were instructed not to take any antipruritic or topical medicine.
  The recruited patients were evaluated and assessed clinically at 2-4-week intervals after treatment by the experienced practitioners who were blinded to the treatment received, in accordance with the criteria described while recruiting the patients.

SECONDARY OUTCOMES:
ADVERSE EFECTS OF DRUGS | 2 weeks
  Skin itching, swelling, and erythema can happen with scabies patients and may exacerbate following permethrin therapy, Mild stinging or burning might occur as a result of the absorption of dead parasite proteins .

CONTACTS AND LOCATIONS:
Overall Officials: Naheed Khan, MBBS, Principal Investigator — Cpsp
Locations (1):
- Combined military hospital, Abbottābād, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ranjkesh MR, Naghili B, Goldust M, Rezaee E. The efficacy of permethrin 5% vs. oral ivermectin for the treatment of scabies. Ann Parasitol. 2013;59(4):189-94. PMID 24791346